CLINICAL TRIAL: NCT05046002
Title: COVID-19 Vaccine-induced Inflammatory Heart Disease Prevalence Registry (COVID-VIHPR)
Brief Title: COVID-19 Vaccine-induced Inflammatory Heart Disease Prevalence Registry
Acronym: COVID-VIHPR
Status: Recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: CTO 3740
Record Dates: First submitted 2021-08-16; First posted 2021-09-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Myocarditis; Pericarditis
MeSH Terms: conditions — Myocarditis; Pericarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — At the time of standard-of-care bloodwork collection, additional research blood samples for biomarker assessment will be collected. Analysis of serum biomarkers such as hs-CRP, ESR, TNF-alpha, IL-1 beta IL-6, and IL-10 may help shed light on the pathway of inflammation. Antibody titres response to mRNA vaccination in younger patients will be of particular interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective (cases): Patients who develop new symptoms of suspected myocarditis/pericarditis within 42 days of receiving a COVID-19 vaccination. The clinical symptoms include chest pain, pressure, or discomfort; dyspnea, shortness of breath, or pain with breathing; palpitations; diaphoresis or sudden death. The symptoms can also be non-specific, including fatigue, abdominal pain, dizziness or syncope, edema, cough or irritability, vomiting, poor feeding, tachypnea or lethargy in young children
- Prospective (Control Negative): Family members/relatives who have been vaccinated in a similar timeframe with the participants but did not experience myocarditis side-effects.
  If a relative is not available, then a voluntary control who has received the same COVID-19 vaccine in a similar time frame can be recruited.
- Retrospective: Identified patients, previously diagnosed with the condition, at participating centers

SUMMARY:
Myocarditis and pericarditis are inflammatory diseases of the myocardium and pericardium, and can be related to different causes, including vaccines. In the past, some people developed inflammatory heart disease after receiving a live or inactive virus vaccine (smallpox vaccine or flu vaccine). Myocarditis was also seen in people with COVID-19. More recently, many countries reported that some people have developed an inflammatory condition of the myocardium or pericardium after receiving a vaccine for COVID-19.

After the COVID-19 vaccination campaigns, doctors have noticed more people presenting to the Emergency Department with chest pain and shortness of breath after receiving the vaccine, symptoms that resemble myocarditis or pericarditis. These symptoms may start between 2 to 10 days following vaccination and are frequently noticed after the second dose of the vaccines. While pericarditis seems to affect people of various age groups and gender, myocarditis is more commonly seen in young males.

The study will consist of two components. 1) The vaccine-induced inflammatory heart disease database will be established. There will be a retrospective chart review looking at vaccine myocarditis/pericarditis (Brighton Criteria Levels 1-3).

2) There will be a prospective, pragmatic design case-control study for vaccine myocarditis/pericarditis. Follow-up telephone interview will be conducted at 6 months, 12 months and yearly up to 4 years. A record search will also be performed at 6 months, 12 months and yearly for 4 years.

The retrospective component of the study will be conducted by identifying patients previously diagnosed with this condition at participating centres.

DETAILED DESCRIPTION:
The study will consist of two components. 1) The vaccine-induced inflammatory heart disease database will be established. There will be a retrospective chart review looking at vaccine myocarditis/pericarditis (Brighton Criteria Levels 1-3).

2) There will be a prospective, pragmatic design case-control study for vaccine myocarditis/pericarditis.

This will be a multi-center study conducted in centers in Canada that treat post-vaccine inflammatory heart disease in both the inpatient and outpatient settings. Patients will be invited to participate in the Registry when they present to the Emergency Department, during inpatient admission, or in the Cardiology Outpatient Clinic. Patients will be invited to ask a relative or friend to contact the research site to serve as controls. The retrospective component of the study will be conducted by identifying patients previously diagnosed with this condition at participating centers.

At some centers, we will collect clinical information and include blood samples for biomarkers at the baseline/recruitment visit and first follow-up visit for cases and at a research study visit for controls. The follow-up visit is expected to be between 4 and 12 weeks after the initial visit.

The UOHI will see the patients for clinical purposes and the research data will be captured at the same time points. These are expected at baseline/initial visit and then a 4-12-weeks follow-up visit. Clinical assessments and bloodwork will be conducted at the two visits. Subsequent follow-up via telephone interview will be conducted after 6 months, 12 months and every year for 4 years, with a script-based questionnaire to ascertain the patient's clinical status and the achievement of clinical endpoints. Patients will be asked to complete a quality-of-life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. All patients eligible for vaccination with a COVID-19 vaccine,
2. At least one cardiac symptom of suspected myocarditis/pericarditis within 42 days of receiving a COVID-19 vaccination. The clinical symptoms include chest pain, pressure, or discomfort; dyspnea, shortness of breath/dyspnea/pain with breathing, palpitations, diaphoresis, syncope, or sudden death.

   OR At least two non-specific symptoms within 42 days of receiving a COVID-19 vaccination. These symptoms include fatigue, abdominal pain, dizziness or syncope, edema, or cough.

   OR No symptoms, but abnormal histopathology or a combination of abnormal cardiac biomarkers with abnormal cardiac imaging (echo or MRI)
3. At least one of the following:

   1. Elevations in Troponin T, Troponin I, or CK-MB (above threshold of normal)
   2. Abnormal MRI (per Brighton Criteria Case Definitions)
   3. Any new or worsening cardiac arrhythmias on ECG or telemetry or Holter monitor (per Brighton Criteria Case Definitions) including those that normalize on recovery.
   4. Abnormal Echocardiographic findings (per Brighton Criteria Case Definitions, see Appendix 2 and 3)
   5. Physical exam finding: Pericardial friction rub or pulsus paradoxus
   6. Pericardial fluid or inflammation by imaging (echo, MRI, or CT) or at least one of the following elevated biomarkers of inflammation: ESR, CRP, hs-CRP, or D-Dimer.
   7. Enlarged heart on chest radiograph.
   8. Histopathologic examination of myocardial tissue (autopsy or endomyocardial biopsy) showed myocardial inflammation

Exclusion Criteria:

1. Clear alternative diagnosis or explanation for the symptoms and findings (e.g. infectious myocarditis such as Lyme carditis). Note: Work-up of alternative diagnosis is dependent on clinical presentation e.g. Lyme carditis (e.g. endemic area, season, bullseye rash) or autoimmune heart disease (e.g. arthritis, rash, recurrence).
2. Symptoms after 42 days of vaccination.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have developed symptoms after receiving a COVID-19 vaccine and meet the inclusion and exclusion criteria are eligible to participate in the registry.
  Family members, vaccinated in a similar timeframe, with similar technology vaccine (e.g. any mRNA) but did not experience myocarditis side-effects - as a negative controls. If a relative is not available, voluntary controls who received the same type of COVID-19 vaccine in a similar time frame can be recruited (friends, roommates) Alternatively, if family members also had similar reactions, they can be recruited as positive controls.
  For the retrospective registry, we would also collect data on COVID-19 myocarditis and pericarditis and all other etiologies of myocarditis or pericarditis.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with autoimmune disease | 30 days
  To identify how many patients (in each group) have a history of autoimmune disease
Composite of MACE | 30 days
  To identify major cardiovascular events - death, ventricular arrhythmia, heart block, heart failure, LV dysfunction (LVEF<55%), cardiac tamponade, re-hospitalization for cardiac reasons

SECONDARY OUTCOMES:
Recurrence of myocarditis/pericarditis | 3 months, 6 months, 12 months, every year for 4 years
  similar symptoms compared to baseline
Atrial arrhythmias | 3 months, 6 months, 12 months, every year for 4 years
  irregular atrial heart rhythms
Cardiovascular mortality | 3 months, 6 months, 12 months, every year for 4 years
  death from any cardiac cause
Quality of life data | 3 months, 6 months, 12 months, every year for 4 years
  EQ-5D-5L questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
To be determined